CLINICAL TRIAL: NCT04231903
Title: Endo-aortic Versus Trans-thoracic Clamping in Right Mini-thoracotomy Mitral Valve Repair: Outcome on Myocardial Pro-tection
Brief Title: Myocardial Protection in Minimally Invasive Mitral Valve Surgery
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Cristina Barbero, MD, PhD, Cardio-thoracic Surgeon, Principal Investigator, University of Turin, Italy
Other Study IDs: 0063123
Record Dates: First submitted 2020-01-05; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Myocardial Protection; Minimally Invasive Surgery; Mitral Valve Prolapse
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EAC: Patients undergoing surgery endo-aortic clamp.
  Interventions: Device: Aortic clamp
- TTC: Patients undergoing surgery through trans-thoracic aortic clamp.
  Interventions: Device: Aortic clamp

INTERVENTIONS:
Device: Aortic clamp — In the firs group an endo-aortic clamp is used and in the second group an external clamp is used.

SUMMARY:
Perfusion strategies and aortic clamping techniques for right mini-thoracotomy mitral valve (MV) surgery have evolved over time and remarkable short- and long-term results have been re-ported. However, some concerns have emerged about the adequacy of myocardial protection dur-ing the minimally invasive approach and about the role of aortic clamping strategies in this contest.

Aim of this study was to compare the efficacy, in terms of myocardial protection, of the en-do-aortic clamp (EAC) versus the trans-thoracic aortic clamp (TTC) in patients undergoing right mini-thoracotomy MV repair.

A single center, prospective observational study was performed between June 2014 to June 2018 on patients undergoing right mini-thoracotomy MV repair with retrograde arterial perfusion and EAC or TTC. The selection of one setting in respect to the other was patient orientated. Myocardial protection was assessed through creatinine kinase-myocardial band (CK-MB) and cardiac Troponin T (cTn-T) blood levels immediately after the surgical procedure and at 6, 12, and 24 hours and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Surgical indication for mitral valve repair.
* Right mini-thoracotomy approach.
* Retrograde arterial perfusion.

Exclusion Criteria:

* Age more than 75 years.
* Cardiac ejection fraction lower than 40%.
* Previous cardiac surgery procedures for coronary artery bypass graft.
* Any degree of coronary artery disease.
* Severe peripheral vascular disease.
* Concomitant procedures for atrial fibrillation ablation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers at our Deparment with diagnosis of mitral valve disease with surgical indication for mitral valve repair through the right mini-thoracotomy approach and retrograde arterial perfusion.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
cTn-T levels immediately after surgery | Immediately after surgery
  Myocardial protection was assessed through cardiac Troponin T (cTn-T) blood levels and compared between the 2 groups of aortic clamping
CK-MB levels immediately after surgery | Immediately after the surgery
  Myocardial protection was assessed through creatinine kinase-myocardial band (CK-MB) blood levels after right mini-thoracotomy mitral valve surgery and compared between the 2 groups of aortic clamping
cTn-T levels 6h | hour 6 after surgery
  Myocardial protection was assessed through cardiac Troponin T (cTn-T) blood levels and compared between the 2 groups of aortic clamping
CK-MB levels 6h | hour 6 after surgery
  Myocardial protection was assessed through creatinine kinase-myocardial band (CK-MB) blood levels after right mini-thoracotomy mitral valve surgery and compared between the 2 groups of aortic clamping
cTn-T levels 12h | hour 12 after surgery
  Myocardial protection was assessed through cardiac Troponin T (cTn-T) blood levels and compared between the 2 groups of aortic clamping
CK-MB levels 12h | hour 12 after surgery
  (CK-MB) blood levels after right mini-thoracotomy mitral valve surgery and compared between the 2 groups of aortic clamping
cTn-T levels 24h | hour 24 after surgery
  Myocardial protection was assessed through cardiac Troponin T (cTn-T) blood levels and compared between the 2 groups of aortic clamping
CK-MB levels 24h | hour 24 after surgery
  Myocardial protection was assessed through cardiac Troponin T (cTn-T) blood levels and compared between the 2 groups of aortic clamping

IPD SHARING:
Plan to Share IPD: Undecided